CLINICAL TRIAL: NCT01371240
Title: Evaluation of Efficiency of Secretin-Assisted Computed Tomography Scan and Secretin-Assisted Magnetic Resonance Imaging in Improving Pancreatic Enhancement and Tumor Conspicuity: Prospective Study
Brief Title: Secretin-Assisted Computed Tomography Scan and Magnetic Resonance Imaging in Improving Pancreatic Tumor Conspicuity
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study never started
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Repligen Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: CC00035
Record Dates: First submitted 2011-06-07; First posted 2011-06-10 (Estimated); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Pancreas Cancer
Keywords: pancreas cancer; MRI; CT scan
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Secretin

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Drug: Secretin Synthetic Human (RG1068) — A maximum dose of 100 consumer unit (CU) of RG1068, synthetic human secretin (Repligen Corporation) or one CU per kg body wt for patients that weight less than 100 kg will be injected (0.2µg of RG1068 are equal to 1CU) (RepliGen Co., Waltham, MA, USA). This dose will be given as an intravenous bolus at 3 minutes before injecting the contrast.

SUMMARY:
Accurate preoperative tumor detection and staging are fundamental for treating patients with pancreatic adenocarcinoma. Patients with unresectable tumors can benefit from being spared an extensive operation associated with substantial morbidity and mortality, cost, and pain. On the other hand, patients with localized disease, which is amenable to surgical removal, have the option of operation. Therefore, accurate staging of pancreatic cancer requires the detection of the tumor, and evaluation of its size, its relationship to major peri-pancreatic vascular structures and portal venous system, locoregional lymph nodes, and distant metastases. Multiple imaging techniques have been used to evaluate the pancreas. Although, at this point, no consensus exists as to the best staging algorithm, multidetector (MD) computed tomogrophy (CT) and Magnetic resonance imaging (MRI) provide sufficient information for the management of most patients.

Patients with a tumor larger than 3 cm are characterized as non-surgical. CT sensitivity in detecting small pancreatic tumors of less than 2 cm is low. Multiple methods have been suggested to increase the sensitivity of CT. The sensitivity of CT increases with using multidetector CT which now has an accuracy rate of about 95-97% for initial detection and approximating that of 100% for staging.

Secretin (a natural hormone produced by the duodenal mucosal cells) is known to increase blood flow to the pancreas. The principal use of secretin in imaging today is in exocrine function of the pancreas or morphological evaluation of the pancreatic duct under ultrasound or MRI. Theoretically, pancreatic contrast enhancement should also increase after secretin administration. This would imply that tumor conspicuity might also be increased if contrast enhancement of the normal pancreas increases. Secretin CT has been advocated by other centers to improve depiction of the ampulla and periampullary/duodenal diseases and to improve contrast enhancement. O'Connell et al, used secretin in patients suspected or with known pancreatic mass and concluded that administration of intravenous secretin leads to greater enhancement of the pancreas with greater tumor conspicuity, than imaging without secretin.

MRI of the pancreas has undergone a major change because it can provide noninvasive images of the pancreatic ducts and the parenchyma. MR cholangiopancreatography (MRCP) enables detection of anatomic variants such as pancreas divisum. Although contrast material-enhanced CT is still considered the gold standard in acute pancreatitis and for the detection of calcifications in chronic pancreatitis, MR imaging and secretin-enhanced MRCP are useful in evaluating pseudocysts and pancreatic disruption.

The role of MR is still debated in pancreatic neoplasms except the cystic lesions where MR imaging provides critical information regarding the lesion's content and a possible communication with the pancreatic ducts. Although some articles have shown that MRI was equivalent to CT in diagnosis and staging, others have shown the opposite. Nishiharu et al. found comparable tumor detection but a benefit with CT, notably for peripancreatic and vascular invasion. Comparing CT, echoendoscopy, and MRI, Soriano et al. demonstrated that CT showed the highest level of precision in primary tumor staging, local-regional staging, vascular invasion, distant metastases, Tumor, node, metastasis (TNM) staging, and tumor resectability. MRI retains its originality in imaging the parenchyma, the pancreatic and biliary ducts, and vascular structures; however, in many institutions, CT remains the reference imaging choice for diagnosing and staging pancreatic cancer. Other than CT's advantages for the tumor, its excellent spatial resolution also provides detailed reconstructions in all planes and arterial mapping and therefore makes it possible to search for surgical contraindications such as celiac trunk stenosis. MRI is still used today as a second-intention tool when there is doubt or when CT and echoendoscopy are not sufficiently conclusive; it is not currently recommended to use MRI in first-intention diagnosis of pancreatic cancer.

The aim of this pilot study is to determine whether the administration of intravenous secretin before contrast-enhanced CT and MRI improves pancreatic enhancement and pancreatic tumor conspicuity and to evaluate which technique is more appropriate for pancreatic tumor detection, staging and evaluation of resectability.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 or above will be included in the study.
2. Patients suspected of pancreatic mass or with a known pancreatic mass would be enrolled in the study.
3. Patients with suspected pancreatic pathology and scheduled for imaging study (CT vs. MRI) will be included if they had obstructive jaundice, with either a stricture in the lower common bile duct on magnetic resonance cholangiopancreatography (MRCP) or a pancreatic mass on ultrasound or other imaging study.

Exclusion Criteria:

1. Patients with known advanced pancreatic tumors and those with previous pancreatic resection will be excluded.
2. Patients with renal insufficiency: increase Cr level or glomerular filteration rate (GFR) of less than 45 ml/min/1.73.
3. Patients who demonstrate increase in Cr level or patients with acute renal injury.
4. Claustrophobic or patients who are not able to tolerate MRI.
5. Patients with previous history of contrast allergies.
6. Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Increase in pancreatic tumor conspicuity. | one year
  Quantitative analysis will be performed using CT attenuation values obtained from the pancreas and from pancreatic tumors. The average CT attenuation will be calculated for the normal pancreatic tissue and any tumor. The mean pancreatic enhancement for the pancreatic and portal venous phases will be obtained by subtracting the mean CT attenuation value on nonenhanced images from the mean CT attenuation obtained from pancreatic and portal venous phase enhanced images. Mean enhancement for the pancreatic and portal venous phases will be calculated for both secretin and nonsecretin patients.
Pancreatic tumor conspicuity on MRI | one year
  The diameter of the main pancreatic duct before and after secretin stimulation will be measured to monitor variations in ductal size.
  The size of the tumor both before secretin administration and afterwards will be measured.

SECONDARY OUTCOMES:
post-injection complications and side effects of secretin | one year
  All patients will be evaluated before the injection and throughout the entire study. Complete physical examination will be performed immediately after the study completion. The patients will be observed for 10 minutes after the study is done and re-evaluated for side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo R Ros, MD MPH PhD, Study Chair — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States